CLINICAL TRIAL: NCT04105543
Title: Therapeutic Combination of CLR 131 With External Beam Radiation in Head and Neck Cancer
Brief Title: CLR 131 Combined With Radiation for Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW19041; P50DE026787 (NIH); 2019-0681 (Other: Institutional Review Board); A534260 (Other: University of Wisconsin - Madison); SMPH/MEDICINE/HEM-ONC (Other: University of Wisconsin - Madison); NCI-2019-05419 (Registry Identifier: NCI Trial ID); Protocol Version 11/9/2021 (Other: UW Madison)
Record Dates: First submitted 2019-09-25; First posted 2019-09-26 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — CLR1404

STUDY DESIGN:
Intervention Model Description: Single center, dose escalation and dose expansion study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CLR 131 Dose Escalation (Experimental): Enrollment will start at dose level 1 (first 4 participants). Participants will receive 2 doses of CLR 131 intravenously with the first dose on day 1 followed by the second dose on day 8.
  Dose Level -1 (de-escalation dose, if toxicities warrant) = 12.5 mCi/m^2 Dose Level 1 (beginning dose) = 15.6 mCi/m^2 Dose Level 2 (escalation dose) = 18.75 mCi/m^2
  Dose escalation will proceed with no limiting toxicities at each level (maximum of 8 participants at each dose level). With maximum tolerated dose confirmed, an expansion phase will proceed.
  Interventions: Drug: CLR 131

INTERVENTIONS:
Drug: CLR 131 — CLR 131 is a radiopharmaceutical dosed intravenously over a period of approximately 30 minutes, dose will be based on total body surface area calculated from actual body weight and height
  Other Names: I-131-CLR1404

SUMMARY:
This is a Phase 1 study of the use of an investigational drug that selectively delivers radiation to malignant tumor cells, CLR 131, in combination with external beam radiation therapy (EBRT) in subjects with locoregionally recurrent head and neck cancer. The trial will enroll up to 12 participants who are amenable to retreatment with radiation therapy. Participants who also have distant metastatic disease may be enrolled on this clinical trial, but they must have evaluable disease that will be clinically treated with radiation therapy, as per standard of care. All participants will receive a dosimetry test dose of CLR 131 to establish drug uptake by the tumor and enable Monte Carlo dose estimation based on CLR 131 SPECT/CT imaging evaluation. Participants showing uptake will receive a cumulative tumor dose of 60-70 Gy using personalized dose calculation (via Monte Carlo methods) of CLR 131 combined with external beam radiation.

DETAILED DESCRIPTION:
Following informed consent, all participants will receive a dosimetry test dose of 15 mCi CLR 131 to establish drug uptake by the tumor and enable Monte Carlo dose estimation based on CLR 131 SPECT/CT imaging evaluation.

Participants who have uptake of the CLR 131 dosimetry test dose at their disease site as determined by the study radiologist will be eligible to participate on the treatment portion of this clinical trial. Participants showing uptake will receive a cumulative tumor dose of 60-70 Gy using personalized dose calculation of CLR 131 (via Monte Carlo) combined with external beam radiation. In this study, we are also studying a subset of up to 6 patients who do not uptake after the CLR 131 test dose, who will still proceed with treatment with CLR 131.

This clinical trial involves two cohorts of subjects: (a) dose escalation and (b) dose expansion. In the dose escalation phase, an mTPI-2 design, an extension of modified toxicity probability interval (mTPI-2), will be used to identify the maximum tolerated dose (MTD) using cohorts of 4 participants and up to 3 dose levels of CLR 131. Participants in the dose escalation phase will receive 2 doses of CLR 131 with the first dose on day 1 followed by the second dose on day 8.

Treatment with CLR 131 on the dose escalation cohort will begin at dose level 1 (15.6 mCi/m2). Participants at dose level 1 will receive an intravenous infusion of CLR 131 at 15.6 mCi/m2 on day 1 followed by a second dose on day 8. Participants at dose level 2 will receive an intravenous infusion of CLR 131 at 18.75 mCi/m2 on day 1 followed by a second dose on day 8.

Once the MTD is determined by the dose escalation phase, participants will be enrolled on the dose expansion cohort. Participants on the dose expansion cohort will receive 2 doses of CLR 131 with the first dose on day 1 followed by the second dose on day 8, with the dose determined by the dose escalation phase.

SPECT/CT imaging will be performed on days 2, 3, 4-6, and 7-8 of the treatment period to visualize and quantitate the biodistribution of CLR 131. Based on these SPECT/CT imaging scans, the Bednarz lab will utilize the Monte Carlo method to predict absorbed dose of CLR 131 to tumors and normal structures.

All participants will start thyroid-protection medication the day prior to the CLR 131 dosimetry test dose and will continue to take thyroid protection medication for 14 days after the last CLR 131 dose.

Based on the calculated absorbed dose of CLR 131 to the specific targeted tissue, the participant will undergo external beam radiation therapy (EBRT) to complete the designated radiation dose outlined in the re-irradiation plan, as per standard of care. Prior to CLR 131 administration and at 3 and 6 months post EBRT, participants will be assessed for changes to swallow function. Prior to CLR 131 administration and at 3, 6 and 12 months post EBRT, quality of life measures and salivary characteristics will be assessed. The investigators anticipate the total study (baseline, CLR 131 administration, EBRT and 3, 6, 12 and 24 month follow up assessments) to take 27 months per participant.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be informed of the investigational nature of the study and must be able to sign a written informed consent.
* Participants with histologically or cytologically confirmed solid malignancy that has recurred in the head and neck (above the clavicles) region, e.g., participants with recurrent cutaneous squamous cell carcinoma, salivary gland tumors or esthesioneuroblastoma are eligible for this clinical trial.
* Participants must have undergone previous curative intent therapy, with radiation as a primary or adjuvant therapy.
* Participants may have distant metastatic disease, as long as the locoregional site of recurrence is deemed eligible for radiation therapy, and treatment of the loco-regional disease is deemed as taking precedence over treatment of the remaining systemic disease.
* Participants must have at least one evaluable (measurable or non-measurable) recurrent lesion that is amenable to radiation therapy.
* Participants must demonstrate uptake of CLR 131 via SPECT/CT imaging, as determined by the study radiologist, in the specified site of recurrent/metastatic disease that is to be treated with radiation therapy. There is a subset of up to 6 patients who may continue with CLR 131 treatment without uptake on the SPECT/CT scan after the test dose.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Participants must have a life expectancy of at least 6 months.
* The participant has adequate hematologic function, as evidenced by:

  * an absolute neutrophil count (ANC) ≥ 1500 / µL
  * hemoglobin ≥9 g/dL (5.58 mmol/L)
  * and platelets ≥100,000 / µL

    * If full-dose anticoagulation therapy is used, platelets ≥ 150,000 / µL are required.

      * If participant is on full-dose anticoagulation therapy, the anticoagulation therapy must be reversible, and reversal of the anticoagulation therapy must not be life-threatening, as judged by the investigator.
* The participant has adequate renal function as defined by:

  * serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or Cockcroft-Gault calculated creatinine clearance >/= 60 ml/min
* The participant has adequate hepatic function as defined by:

  * total bilirubin ≤ 1.5 mg/dL (25.65 μmol/L)
  * aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the ULN
* Women of childbearing potential (WOCP) have a confirmed negative urine pregnancy test within 24 hours prior to test dose of CLR 131.
* Participants must use a medically acceptable method of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence during the study participation and for 6 months after last dose of study drug. Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
* Men who are not surgically or medically sterile agree to use an acceptable method of contraception. Male participants with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must abstain from intercourse for three weeks after each CLR 131 dose and agree to use condoms at least 6 months after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.

Exclusion Criteria:

* Recurrent tumor recommended for surgical resection based on multidisciplinary Head and Neck Oncology Tumor Board Review
* Thyroid cancer
* Known hypersensitivity to iodine
* Other concurrent severe and/or uncontrolled concomitant medical or psychiatric conditions (e.g. active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol, per investigator discretion
* Chemotherapy or major surgery within 4 weeks, or radiotherapy within 2 weeks prior to test dose of CLR 131.
* Participants with clinically significant adverse events due to agents administered more than 4 weeks prior to test dose of CLR 131 (alopecia and fatigue excluded). Clinical significance to be determined by investigator.
* The participant is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment.
* Any ongoing or active infection, including active tuberculosis, hepatitis B or C, or known infection with the human immunodeficiency virus (HIV)
* Concurrent treatment with any other anti-cancer or investigational agents. Participants cannot be receiving concomitant chemotherapy, radiotherapy, experimental therapy or any other therapy not otherwise outlined by the trial for the purposes of anti-cancer treatment.
* Participants with a history of or concurrent second primary malignancy (stage III or IV) within 5 years to study enrollment are excluded.
* Participants with a history of prior invasive malignancy (except early-stage I or II non-melanomatous skin cancer, carcinoma in situ of the breast, cervical carcinoma in situ, stage I-II papillary thyroid cancer, or low or very low-risk prostate cancer which has been completely treated with surgery or radiation) treated within 2 years of study enrollment are excluded.
* Participants that have had total body or hemibody irradiation, or have had prior systemic radioisotope therapy (except for benign thyroid disease)
* Poor venous access and will be unable to receive study drug into a peripheral venous catheter.
* Significant traumatic injury within 6 weeks prior to enrollment
* Extradural tumor in contact with the spinal cord or tumor located where swelling in response to therapy may impinge upon the spinal cord
* Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
* History of myocardial infarction, ventricular arrhythmia, stable/unstable angina, symptomatic congestive heart failure, coronary/peripheral artery bypass graft or stenting or other significant cardiac disease within 6 months prior to study entry
* QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥480 ms.
* Any condition requiring the use of immunosuppression, excluding rheumatologic conditions treated with stable doses of corticosteroids (equivalent to £ prednisone 10 mg daily)
* Ongoing hemodialysis or peritoneal dialysis
* Poorly controlled severe Chronic Obstructive Pulmonary Disease (COPD)
* Uncontrolled hypothyroidism or hyperthyroidism
* Any medical condition that predisposes the subject to uncontrolled bleeding such as hemophilia, factor deficiencies, severe liver disease, or von Willebrand disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justine Bruce, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruce JY, Burr A, Kimple RJ, Adam DP, Yu M, Piaskowski SM, Glazer TA, Hill P, Hartig GK, McCulloch TM, Wieland AM, Trask D, Oliver K, Longcor J, Rogus-Pulia N, Cho SY, Bednarz B, Harari PM. Safety and toxicity of Iopofosine I 131 (CLR 131) with external beam radiation therapy in recurrent or metastatic head and neck cancer: results of a phase 1 single-centre, open-label, single-arm, dose escalation and dose expansion study. EBioMedicine. 2025 Jan;111:105496. doi: 10.1016/j.ebiom.2024.105496. Epub 2024 Dec 12. PMID 39671752
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from October 2020 to February 2022 at the UW Hospital and Clinics.
Groups:
- CLR 131 Dose Escalation: Enrollment will start at dose level 1 (first 4 participants). Participants will receive 2 doses of CLR 131 intravenously with the first dose on day 1 followed by the second dose on day 8.
  Dose Level -1 (de-escalation dose, if toxicities warrant) = 12.5 mCi/m^2 Dose Level 1 (beginning dose) = 15.6 mCi/m^2 Dose Level 2 (escalation dose) = 18.75 mCi/m^2
  Dose escalation will proceed with no limiting toxicities at each level (maximum of 8 participants at each dose level). With maximum tolerated dose confirmed, an expansion phase will proceed.
  CLR 131: CLR 131 is a radiopharmaceutical dosed intravenously over a period of approximately 30 minutes, dose will be based on total body surface area calculated from actual body weight and height
Period: CLR Dose Level 1: 15.6mCi
Arm/Group | CLR 131 Dose Escalation
Started | 4
Participants With Dose Limiting Toxicities | 1
Completed | 4
Not Completed | 0
Period: Dose Held at Dose Level 1: 15.6mCi
Arm/Group | CLR 131 Dose Escalation
Started (Investigators held dose at 15.6mCi as 1 participant had a dose limiting toxicity. N=12 includes the 4 participants initially enrolled into this dose level.) | 12
Completed Treatment | 12
Primary Analysis Population | 12
Overall Response Rate Analysis Population | 11
Completed Baseline Salivary Measures | 10
Completed 3 Months Post EBRT Salivary Measures | 9
Completed 6 Months Post EBRT Salivary Measures | 5
Completed 12 Months Post EBRT QoL Measures | 0
Died While on Study | 8
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- CLR 131 Dose Escalation: Enrollment will start at dose level 1 (first 4 participants). Participants will receive 2 doses of CLR 131 intravenously with the first dose on day 1 followed by the second dose on day 8.
  Dose Level -1 (de-escalation dose, if toxicities warrant) = 12.5 mCi/m^2 Dose Level 1 (beginning dose) = 15.6 mCi/m^2 Dose Level 2 (escalation dose) = 18.75 mCi/m^2
  Dose escalation will proceed with no limiting toxicities at each level (maximum of 8 participants at each dose level). With maximum tolerated dose confirmed, an expansion phase will proceed.
  CLR 131 is a radiopharmaceutical dosed intravenously over a period of approximately 30 minutes, dose will be based on total body surface area calculated from actual body weight and height
Arm/Group | CLR 131 Dose Escalation
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 65.5 [47 to 84]
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 2
  50-59 years | 3
  60-69 years | 2
  70-79 years | 3
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status of 0 means "Fully active, able to carry on all pre-disease performance without restriction", 1 means "Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work" (from ECOG-ACRIN website)
  Participants
    ECOG 0 | 9
    ECOG 1 | 3
Primary Tumor Site [Count of Participants; unit: Participants]
  Oropharynx | 5
  Nasopharynx | 1
  Larynx | 1
  Oral cavity | 4
  Salivary Gland | 1
T stage [Count of Participants; unit: Participants] — Primary Tumor Stage (T stage), T1 and T2 are less than or equal to 5 cm and T3 and T4 are greater than 5 cm
  Participants
    T1 and T2 | 6
    T3 and T4 | 6
N stage [Count of Participants; unit: Participants] — Nodal involvement (N stage), N0 - N3, where N0 is no metastasis and N3 is higher levels of metastasis.
  Participants
    N0 and N1 | 6
    N2 and N3 | 6
AJCC 8th ed. stage [Count of Participants; unit: Participants] — American Joint Commission on Cancer (AJCC) cancer staging scheme that combines primary tumor stage, nodal involvement, and metastasis. Stage I would be the most localized and Stage IV would be the most regional. Stage IV laryngeal cancer is further divided: Stage IVA is advanced local/regional disease and Stage IVB is advanced distant metastatic disease.
  Participants
    Stage I | 2
    Stage II | 3
    Stage III | 3
    Stage IVA | 2
    Stage IVB | 2
Initial Treatment at Diagnosis [Count of Participants; unit: Participants]
  Surgical Resection: No adjuvant treatment | 1
  Surgical Resection: Adjuvant radiation | 4
  Surgical Resection: Adjuvant chemoradiation | 2
  Definitive Chemoradiation | 5
Recurrence Status at Study Entry [Count of Participants; unit: Participants]
  First Recurrence | 6
  Multiply Recurrent | 6
  Metastatic Disease | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Related Adverse Events
Description: Incidence of adverse events assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Adverse Events Grading (1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death)
Time Frame: up to 18 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1: Grade 1 Treatment (CLR 131) Related Adverse Events
- Grade 2: Grade 2 Treatment (CLR 131) Related Adverse Events
- Grade 3: Grade 3 Treatment (CLR 131) Related Adverse Events
- Grade 4: Grade 4 Treatment (CLR 131) Related Adverse Events
Arm/Group | Grade 1 | Grade 2 | Grade 3 | Grade 4
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Blood and lymphatic system disorders: Anemia | 4 | 2 | 4 | 1
  Blood and lymphatic system disorders: Febrile neutropenia | 0 | 0 | 2 | 0
  Gastrointestinal disorders: Dry mouth | 2 | 1 | 0 | 0
  Gastrointestinal disorders: Dysphagia | 0 | 2 | 0 | 0
  Gastrointestinal disorders: Mucositis oral | 1 | 0 | 1 | 0
  Gastrointestinal disorders: Nausea | 0 | 1 | 0 | 0
  Gastrointestinal disorders: Salivary Duct Inflammation | 1 | 0 | 0 | 0
  General disorders: Fatigue | 4 | 2 | 0 | 0
  General disorders: Fever | 1 | 0 | 0 | 0
  General disorders: Pain | 0 | 1 | 0 | 0
  Infections and infestations: Thrush | 0 | 1 | 0 | 0
  Injury, poisoning and procedural complications: Dermatitis Radiation | 1 | 0 | 0 | 0
  Investigations: Lymphocyte count decreased | 0 | 0 | 5 | 4
  Investigations: Neutrophil count decreased | 0 | 1 | 1 | 7
  Investigations: Platelet count decreased | 1 | 1 | 3 | 6
  Investigations: Thyroid stimulating hormone increased | 1 | 0 | 0 | 0
  Investigations: Weight loss | 0 | 2 | 0 | 0
  Investigations: White blood cell decreased | 0 | 2 | 2 | 7
  Metabolism and nutrition disorders: Anorexia | 1 | 1 | 0 | 0
  Musculoskeletal and connective tissue disorders: Fibrosis deep connective tissue | 1 | 0 | 0 | 0
  Nervous system disorders: Dysgeusia | 1 | 0 | 0 | 0
  Nervous system disorders: Headache | 1 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: Oropharyngeal pain | 2 | 0 | 0 | 0

2. Primary Outcome: Summary of Adverse Events Possibly Related to Treatment
Description: Adverse Events Grading (1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death)
Time Frame: up to 18 weeks
Measure: Count of Participants; unit: Participants
Groups:
- All Adverse Events: All Adverse Events that are Possibly Related to Treatment
- Adverse Events Greater Than or Equal to Grade 3: Adverse Events greater than or equal to grade 3 that are Possibly Related to Treatment.
Arm/Group | All Adverse Events | Adverse Events Greater Than or Equal to Grade 3
Number analyzed (Participants) | 12 | 12
Participants
  Thrombocytopenia | 11 | 9
  Leukopenia | 11 | 9
  Lymphopenia | 9 | 9
  Neutropenia | 9 | 8
  Anemia | 11 | 5
  Fatigue | 6 | 0
  Dry mouth | 3 | 0
  Pain, Oral and Oropharyngeal | 3 | 0
  Febrile neutropenia | 2 | 2
  Mucositis oral | 2 | 1
  Anorexia | 2 | 0
  Dysphagia | 2 | 0
  Weight loss | 2 | 0

3. Secondary Outcome: CLR 131 Tumor Uptake Via SPECT/CT Imaging
Description: Investigators will use SPECT/CT imaging scans to predict the adsorbed dose of CLR 131 to tumors with the Monte Carlo method.
Time Frame: Up to 8 days
Measure: Mean (Full Range); unit: gray (Gy)
Groups:
- CLR 131: Participants will receive 2 doses of CLR 131 intravenously with the first dose on day 1 followed by the second dose on day 8.
  Dose Level = 15.6 mCi/m^2
  CLR 131 is a radiopharmaceutical dosed intravenously over a period of approximately 30 minutes, dose will be based on total body surface area calculated from actual body weight and height
Arm/Group | CLR 131
Number analyzed (Participants) | 12
gray (Gy) | 6.23 [2.65 to 8.69]

4. Secondary Outcome: Median Radiation Treatment Time
Time Frame: up to 14 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | CLR 131
Number analyzed (Participants) | 12
days | 43 [36 to 44]

5. Secondary Outcome: Number of Dose Delays
Time Frame: up to 14 weeks
Measure: Count of Units; unit: doses
Units Other Than Participants: doses
Arm/Group | CLR 131
Number analyzed (Participants) | 12
Number analyzed (doses) | 24
doses
  Due to Toxicity | 0
  Due to Production Difficulties | 1

6. Secondary Outcome: Response Rates
Description: Complete response (CR), disappearance of all tumors; Partial response (PR), at least 30% decrease in the sum of the longest diameter of target tumors; Stable disease (SD), no increase or decrease to tumor size; Progressive disease (PD), increasing tumor size. RECIST v1.1, Response Evaluation Criteria in Solid Tumors version 1.
Time Frame: 6 months post completion of EBRT, up to 9 months on study
Population: One Participant did not undergo post treatment cross-sectional imaging and thus did not have any response data.
Measure: Count of Participants; unit: Participants
Arm/Group | CLR 131
Number analyzed (Participants) | 11
Participants
  Complete Response | 7
  Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 2

7. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR defined as the proportion of subjects who experience either a partial response or complete response within 6 months post completion of EBRT as measured by standard of care imaging (e.g. CT, MR, PET-MR).
Time Frame: 6 months post completion of EBRT, up to 9 months on study
Population: One Participant did not undergo post treatment cross-sectional imaging and thus did not have any response data.
Measure: Count of Participants; unit: Participants
Arm/Group | CLR 131
Number analyzed (Participants) | 11
Participants | 8

8. Secondary Outcome: Swallow Function: DIGEST Scale
Description: Swallow function assessed by Dynamic Imaging Grade of Swallowing Toxicity (DIGEST) scale before and after treatment. The DIGEST scale cross references a clinician determined 'safety' grade with an 'efficiency' grade for an overall score between 0-4 where 0 is asymptomatic and 4 is life threatening. Data collected at baseline, 3 months, and 6 months post completion of external beam radiation therapy (EBRT).
Time Frame: up to 6 months post completion of EBRT (up to 9 months on study)
Population: Unable to collect data from all participants at all timepoints
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- DIGEST Overall Grade: The Overall Grade combines the safety and efficacy scores as a measure of pharyngeal dysphagia, generally 0 is asymptomatic to 4 is life-threatening, specifically:
  * 0 (no pharyngeal dysphagia)
  * 1 (mild pharyngeal dysphagia)
  * 2 (moderate pharyngeal dysphagia)
  * 3 (severe pharyngeal dysphagia)
  * 4 (life-threatening pharyngeal dysphagia)
- DIGEST Safety Grade: Safety measures the impairment when swallowing related to aspiration, generally 0 is asymptomatic to 4 is life-threatening, specifically:
  * 0 (no impairment)
  * 1 (mild impairment)
  * 2 (moderate impairment)
  * 3 (severe impairment)
  * 4 (life-threatening impairment)
- DIGEST Efficacy Grade: Efficacy Measures the impairment related to type of bolus swallowed, generally 0 is asymptomatic to 4 is life-threatening, specifically:
  * 0 (minimal to no residue)
  * 1 (less than half residue)
  * 2 (majority residue, solid bolus types; 50-90%)
  * 3 (majority residue; liquid bolus type; 50-90%)
  * 4 (near complete residue, >90%)
Arm/Group | DIGEST Overall Grade | DIGEST Safety Grade | DIGEST Efficacy Grade
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  baseline | 2 (1.075) | 1 (0.9428) | 3 (1.633)
  3 months post EBRT: number analyzed (Participants) | 9 | 9 | 9
  3 months post EBRT | 2 (1.30) | 1 (0.928) | 3 (1.58)
  6 months post EBRT: number analyzed (Participants) | 5 | 5 | 5
  6 months post EBRT | 3 (1.3) | 2 (1.14) | 3 (1.34)

9. Secondary Outcome: Quality of Life: MDADI Score
Description: Quality of life assessed by MD Anderson Dysphagia Inventory score (MDADI) before and after treatment. MDADI is a 36-item self-assessment with global, emotional, functional, and physical sub-scales. Total possible composite score range is 20-100 where 20 is extremely low functioning and 100 is high functioning. Data collected at baseline, 3 months, and 6 months, and 12 months post EBRT.
Time Frame: Assessed at 3 months and 6 months post EBRT (6 months and 9 months post-baseline). Originally pre-specified to be assessed at 12 months post EBRT, data not collected
Population: Unable to collect data from all participants at all timepoints
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | CLR 131
Number analyzed (Participants) | 10
score on a scale
  baseline | 71.6 (15.9)
  3 months post EBRT: number analyzed (Participants) | 9
  3 months post EBRT | 62.1 (20.6)
  6 months post EBRT: number analyzed (Participants) | 5
  6 months post EBRT | 55.8 (7.68)
  12 months post EBRT: number analyzed (Participants) | 0
Statistical Analysis 1: Comparison: CLR 131; Wilcoxon Signed Rank Tests for MDADI Composite Baseline to 3 months (n=9); Test type: Other — nonparametric rank test; p = 0.173, Wilcoxon Signed Rank Tests; Median Difference (Final Values) = -4.22, 95% CI 2-sided [-12.64 to 4.24]
Statistical Analysis 2: Comparison: CLR 131; Wilcoxon Signed Rank Test for MDADI Composite Baseline to 6 months (n=5); Test type: Other — nonparametric rank test; p = 0.225, Wilcoxon Signed Rank Test; Median Difference (Final Values) = -9.998, 95% CI 2-sided [-28.43 to 7.39]

10. Secondary Outcome: Stimulated Salivary Flow
Description: Stimulated Salivary Flow before and after treatment (mL/min). Data collected at baseline, 3 months, and 6 months post EBRT.
Time Frame: up to 6 months post completion of EBRT (up to 9 months on study)
Population: Unable to collect data from all participants at all timepoints
Measure: Median (Standard Deviation); unit: ml/min
Arm/Group | CLR 131
Number analyzed (Participants) | 9
ml/min
  baseline | 0.24 (0.26)
  3 months post EBRT: number analyzed (Participants) | 8
  3 months post EBRT | 0.18 (0.10)
  6 months post EBRT: number analyzed (Participants) | 4
  6 months post EBRT | 0.21 (0.21)
Statistical Analysis 1: Comparison: CLR 131; Wilcoxon Signed Rank Tests for Stimulated Saliva Flow Baseline to 3 months (n=8); Test type: Other — nonparametric rank test; p = 0.779, Wilcoxon Signed Rank Tests; Median Difference (Final Values) = -0.037, 95% CI 2-sided [-0.246 to 0.09]
Statistical Analysis 2: Comparison: CLR 131; Wilcoxon Signed Rank Test for Stimulated Saliva Flow Baseline to 6 months (n=4); Test type: Other — nonparametric rank test; p = 0.465, Wilcoxon Signed Rank Test; Median Difference (Final Values) = -0.049, 95% CI 2-sided [-0.218 to 0.12]

11. Secondary Outcome: EORTC QLQ-C30 Scores
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is a 30-item instrument measures quality of life in cancer patients. It is scored from 0-100 where higher scores indicate higher level of response in function, symptomatology, or global health.
Time Frame: up to 6 months post completion of EBRT (up to 9 months on study)
Population: Unable to collect data from all participants at all timepoints
Measure: Median (Standard Deviation); unit: score on a scale
Groups:
- EORTC QLQ-C30 Functional Scores: EORTC QLQ-C30 Functional Scores range from 0-100, higher scores indicate higher level of response (higher functioning).
- EORTC QLQ-C30 Symptom Scores: EORTC QLQ-C30 Symptom Scores range from 0-100, higher scores indicate higher level of response (higher symptomatology)
- EORTC QLQ-C30 Global Health Status Scores: EORTC QLQ-C30 Global Health Status Scores range from 0-100, higher scores indicate higher level of response (higher global health).
Arm/Group | EORTC QLQ-C30 Functional Scores | EORTC QLQ-C30 Symptom Scores | EORTC QLQ-C30 Global Health Status Scores
Number analyzed (Participants) | 10 | 10 | 10
score on a scale
  baseline | 76.7 (16.7) | 23.08 (17.92) | 50 (13.82)
  3 months post EBRT: number analyzed (Participants) | 9 | 9 | 9
  3 months post EBRT | 72.2 (13.1) | 26.92 (12.28) | 54.2 (19.32)
  6 months post EBRT: number analyzed (Participants) | 5 | 5 | 5
  6 months post EBRT | 71.1 (11.2) | 28.21 (19.39) | 58.3 (15.59)
Statistical Analysis 1: Comparison: EORTC QLQ-C30 Functional Scores; Wilcoxon Signed Rank Tests for EORTC QLQ-C30 Functional Score Baseline to 3 months (n=9); Test type: Other — nonparametric rank test; p = 0.213, Wilcoxon Signed Rank Tests; Median Difference (Final Values) = -4.444, 95% CI 2-sided [-14.4 to 4.4]
Statistical Analysis 2: Comparison: EORTC QLQ-C30 Functional Scores; Wilcoxon Signed Rank Test for EORTC QLQ-C30 Functional Scores Baseline to 6 months (n=5); Test type: Other — nonparametric rank test; p = 0.686, Wilcoxon Signed Rank Test; Median Difference (Final Values) = -6.667, 95% CI 2-sided [-17.8 to 20]
Statistical Analysis 3: Comparison: EORTC QLQ-C30 Symptom Scores; Wilcoxon Signed Rank Tests for EORTC QLQ-C30 Symptom Score Baseline to 3 months (n=9); Test type: Other — nonparametric rank test; p = 0.498, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 3.846, 95% CI 2-sided [-0.769 to 12.82]
Statistical Analysis 4: Comparison: EORTC QLQ-C30 Symptom Scores; Wilcoxon Signed Rank Test for EORTC QLQ-C30 Symptom Scores Baseline to 6 months (n=5); Test type: Other — nonparametric rank test; p = 0.416, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 10.256, 95% CI 2-sided [-15.39 to 35.89]
Statistical Analysis 5: Comparison: EORTC QLQ-C30 Global Health Status Scores; Wilcoxon Signed Rank Tests for EORTC QLQ-C30 Global Health Status Score Baseline to 3 months (n=9); Test type: Other — nonparametric rank test; p = 0.778, Wilcoxon Signed Rank Test; Median Difference (Final Values) = -8.33, 95% CI 2-sided [-20.84 to 16.67]
Statistical Analysis 6: Comparison: EORTC QLQ-C30 Global Health Status Scores; Wilcoxon Signed Rank Test for EORTC QLQ-C30 Global Health Status Scores Baseline to 6 months (n=5); Test type: Other — nonparametric rank test; p = 0.89, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 0, 95% CI 2-sided [-25 to 25]

12. Secondary Outcome: Xerostomia Quality-of-Life Scale (XeQoLS) Scores
Description: The XeQoLS questionnaire measures the effects of xerostomia on oral health-related quality of life. The questionnaire consists of 15 items, each rated on a 0-to-4 point Likert scale, for a total possible range of scores from 0 to 60, with higher scores indicating more severe symptom burden.
Time Frame: up to 6 months post completion of EBRT (up to 9 months on study)
Population: Unable to collect data from all participants at all timepoints
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | CLR 131
Number analyzed (Participants) | 10
score on a scale
  baseline | 15 (14.4)
  3 months post EBRT: number analyzed (Participants) | 9
  3 months post EBRT | 16.5 (16.9)
  6 months post EBRT: number analyzed (Participants) | 5
  6 months post EBRT | 18 (13.1)
Statistical Analysis 1: Comparison: CLR 131; Wilcoxon Signed Rank Tests for XeQOL Baseline to 3 months (n=9); Test type: Other — nonparametric rank test; p = 0.138, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 3.5, 95% CI 2-sided [-2 to 9.5]
Statistical Analysis 2: Comparison: CLR 131; Wilcoxon Signed Rank Test for XeQOL Baseline to 6 months (n=5); Test type: Other — nonparametric rank test; p = 0.225, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 6, 95% CI 2-sided [-10 to 16]

13. Secondary Outcome: Xerostomia Inventory Score
Description: The Xerostomia Inventory is an 11-item survey scored on a 5 point-likert scale (never, hardly ever, occasionally, fairly often, very much). Total possible range of scores is from 11-55, with higher scores indicating increased mouth dryness.
Time Frame: up to 6 months post completion of EBRT (up to 9 months on study)
Population: Unable to collect data from all participants at all timepoints
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | CLR 131
Number analyzed (Participants) | 10
score on a scale
  baseline | 34.5 (9.38)
  3 months post EBRT: number analyzed (Participants) | 9
  3 months post EBRT | 34.5 (10.75)
  6 months post EBRT: number analyzed (Participants) | 5
  6 months post EBRT | 36.0 (8.08)
Statistical Analysis 1: Comparison: CLR 131; Wilcoxon Signed Rank Tests for Xerostomia Inventory Baseline to 3 months (n=9); Test type: Other — nonparametric rank test; p = 0.674, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 0.500, 95% CI 2-sided [-3 to 5]
Statistical Analysis 2: Comparison: CLR 131; Wilcoxon Signed Rank Test for Xerostomia Inventory Baseline to 6 months (n=5); Test type: Other — nonparametric rank test; p = 0.892, Wilcoxon Signed Rank Test; Median Difference (Final Values) = 0, 95% CI 2-sided [-6 to 6]

ADVERSE EVENTS:
Time Frame: up to 85 days
Description: SAEs through 85 days post first treatment of CLR131 reported regardless of attribution. After day 85, SAE's that had an attribution of at least possibly would be collected and reported.
  AEs will be recorded from time of informed consent until 28 days after last EBRT treatment or 85 days after first treatment dose of CLR 131, whichever is later. AEs will be recorded whether they are considered related to the study drug(s). Xerostomia Inventory Score was not an instrument to collect AE data
Arm/Group | CLR 131 Dose Escalation
All-Cause Mortality (participants affected / at risk) | 8/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLR 131 Dose Escalation (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Failure to thrive
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Neck
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pneumonia
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLR 131 Dose Escalation (N=12)
Anemia (Blood and lymphatic system disorders) | 10 (10)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (8)
Fever (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Mucosal infection (Infections and infestations) | 2 (2)
Thrush (Infections and infestations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 (6)
Lymphocyte count decreased (Investigations) | 10 (10)
Neutrophil count decreased (Investigations) | 10 (10)
Platelet count decreased (Investigations) | 9 (9)
Thyroid stimulating hormone increased (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Neuralgia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oral Pharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Lymphedema (Vascular disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT04105543/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT04105543/ICF_001.pdf